CLINICAL TRIAL: NCT07159412
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Huazhi Rougan Granule Combined With High-Dose Dual Therapy for Helicobacter Pylori Infection Complicated With Metabolic-associated Steatohepatitis (Dampness-Heat Accumulation Syndrome)
Brief Title: Huazhi Rougan Granule as an Add-On Therapy for H. Pylori Infection With Metabolic-associated Steatohepatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20250819-12
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Helicobacter Pylori Infection; Metabolic-associated Steatohepatitis; High-dose Dual Therapy; Huazhi Rougan Granule

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Drug: Vonoprazan-amoxicillin combined with Huazhi Rougan Granule
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Vonoprazan-amoxicillin combined with Huazhi Rougan Granule placebo

INTERVENTIONS:
Drug: Vonoprazan-amoxicillin combined with Huazhi Rougan Granule — Vonoprazan-amoxicillin dual therapy combined with Huazhi Rougan Granule
  Arms: Intervention Group
Drug: Vonoprazan-amoxicillin combined with Huazhi Rougan Granule placebo — Vonoprazan-amoxicillin dual therapy combined with Huazhi Rougan Granule placebo
  Arms: Placebo Group

SUMMARY:
This study employed a double-blind, randomized, placebo-controlled design. Eligible treatment-naïve patients with Helicobacter pylori (Hp) infection complicated by metabolic-associated steatohepatitis (MASH) (dampness-heat accumulation syndrome) were enrolled and randomly assigned to either the experimental group or the placebo control group. Both groups received a 2-week Hp eradication regimen consisting of vonoprazan (20 mg twice daily) and amoxicillin (1000 mg three times daily). The experimental group additionally received active Huazhi Rougan Granule (taken orally three times daily, one sachet each time, with a 6-day medication followed by a 1-day drug holiday per cycle), while the placebo control group received an identical matching placebo on the same schedule. The study aims to evaluate the synergistic therapeutic efficacy of Huazhi Rougan Granule in combination with the vonoprazan-amoxicillin dual therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years;
2. Meeting the diagnostic criteria for metabolic-associated steatohepatitis (MASH) and the traditional Chinese medicine syndrome differentiation criteria for dampness-heat accumulation pattern;
3. Initial treatment for H. pylori infection (positive 13C- or 14C-urea breath test);
4. Signed informed consent form.

Exclusion Criteria:

1. Individuals with fatty liver caused by chronic heart failure, malnutrition, or pregnancy; those with fatty liver syndrome in encephalopathy, abetalipoproteinemia, or localized fatty liver;
2. Patients with severe fatty liver accompanied by ascites, edema, hyponatremia, hypokalemia, or other signs suggestive of cirrhosis; those with hepatitis or cirrhosis caused by viruses, drug toxicity, autoimmune diseases, or other factors;
3. Individuals using hepatoprotective, enzyme-lowering, or lipid-lowering medications that may interfere with efficacy evaluation;
4. Pregnant or lactating women;
5. Patients with severe primary cardiovascular, renal, or other life-threatening diseases;
6. Individuals with a history of cancer;
7. Those positive for HCV antibody, HIV antibody, or HBsAg with detectable HBV-DNA levels;
8. Individuals with a history of alcohol abuse (≥210 g/week for males or ≥140 g/week for females) or substance abuse;
9. Those with known hypersensitivity to any component of the study drug;
10. Participation in another clinical trial within 3 months prior to screening;
11. Use of Chinese herbal medicines for the treatment of non-alcoholic simple fatty liver within 2 weeks prior to screening;
12. Individuals deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | At the end of the 12-week treatment period.
  Patients must undergo a follow-up 13C-urea breath test (13C-UBT) after treatment completion to determine eradication success. A DOB value < 4‱ is considered indicative of successful eradication. The eradication rate is calculated as follows: (number of successfully eradicated patients in each group / total number of patients in that group) × 100.00%.

IPD SHARING:
Plan to Share IPD: No